CLINICAL TRIAL: NCT07301983
Title: Evaluation of Lymph Node Analysis Using One Step Nucleic Acid Amplification (OSNA) in Patients With Lung Cancer Who Underwent Robotic Lung Resection, Comparison With Traditional Methods
Acronym: LALC
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Gaetano Romano, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 22283
Record Dates: First submitted 2025-11-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; early-stage NSCLC; robotic surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients: patients with no other cancer affected by early stage NSCLC
  Interventions: Diagnostic Test: lymph node analysis using the OSNA assay

INTERVENTIONS:
Diagnostic Test: lymph node analysis using the OSNA assay — lymph node analysis using the OSNA assay in early stage NSCLC patients

SUMMARY:
This prospective study aims to evaluate the effectiveness of the One-Step Nucleic Acid Amplification (OSNA) technique for detecting micrometastases in lymph nodes of patients with clinical stage I-II non-small cell lung cancer (NSCLC) undergoing robotic lung resection. OSNA targets CK19 mRNA expression in order to improve the accuracy of mediastinal lymph node staging. The secondary objectives are to identify skip metastases, evaluate the potential for pathological upstaging and analyse long-term outcomes such as overall survival (OS) and disease-free survival (DFS).

This prospective study was approved by the local Ethics Committee in December 2022, and patient enrolment began in May 2023. The inclusion criteria were:

* Resectable non-small cell lung cancer (NSCLC).
* Clinical stage I-II.
* Absence of pathological lymphadenopathy in preoperative staging (cN0). The exclusion criteria included:
* Clinically advanced NSCLC
* Neoadjuvant chemo-immunotherapy
* Presence of other oncological diseases
* Patient refusal to participate. All patients underwent robotic anatomical lung resection combined with systematic lymphadenectomy. Patients were randomised into two groups based on the lymph node (LN) analysis method: OSNA technique or standard histopathological analysis (hematoxylin and eosin or immunohistochemistry).

DETAILED DESCRIPTION:
This prospective study aims to evaluate the effectiveness of the One-Step Nucleic Acid Amplification (OSNA) technique for detecting micrometastases in lymph nodes of patients with clinical stage I-II non-small cell lung cancer (NSCLC) undergoing robotic lung resection. OSNA targets CK19 mRNA expression in order to improve the accuracy of mediastinal lymph node staging.

Cytokeratin 19 is a cytoskeletal component exclusively found in normal or neoplastic epithelial cells, and its presence in lymph nodes serves as an indicator of involvement by tumor cells of epithelial origin.The OSNA method represents a novel approach that determines the number of mRNA copies in the homogenized entire lymph node, overcoming the limitations of hematoxylin- eosin and immunohistochemistry methods that only analyze histological sections and avoiding sampling bias due to the non-uniform localization of metastatic foci. The present study aims to evaluate the advantages of using molecular lymph node assessment in homogeneous samples of patients with the same clinical stage of tumour presentation, stage I and II N0 NSCLC, to optimise data comparison and reduce the risk of potential bias.

Secondary objectives will be the identification of skip metastases and lymph node upstaging.

The future perspective of the study is to analyse long-term follow-up data through outpatient surveillance and radiological examinations to estimate possible disease recurrence and mortality rates in patients The secondary objectives are to identify skip metastases, evaluate the potential for pathological upstaging and analyse long-term outcomes such as overall survival (OS) and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* Resectable non-small cell lung cancer (NSCLC)
* Clinical stage I-II
* Absence of pathological lymphadenopathy in preoperative staging (cN0)

Exclusion Criteria:

* Clinically advanced NSCLC
* Prior neoadjuvant chemo-immunotherapy
* Presence of other oncological diseases
* Patient refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with clinical stage I-II non-small cell lung cancer (NSCLC) undergoing robotic lung resection.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with nodal micrometastasis with OSNA analisis | through study completion, an average of 5 year
  The primary aim of this prospective study is to assess the effectiveness of the One- Step Nucleic Acid Amplification (OSNA) technique in detecting lymph node micrometastases in patients with clinical stage I-II non-small cell lung cancer (NSCLC) undergoing robotic lung resection. By targeting CK19 mRNA expression, OSNA aims to improve the accuracy of mediastinal lymph node staging.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Haustein UF. Pemphigus vulgaris in association with silicosis. Eur J Dermatol. 2000 Dec;10(8):614-6. PMID 11125324
- [Background] Nakagawa K, Asamura H, Tsuta K, Nagai K, Yamada E, Ishii G, Mitsudomi T, Ito A, Higashiyama M, Tomita Y, Inoue M, Morii E, Matsuura N, Okumura M. The novel one-step nucleic acid amplification (OSNA) assay for the diagnosis of lymph node metastasis in patients with non-small cell lung cancer (NSCLC): Results of a multicenter prospective study. Lung Cancer. 2016 Jul;97:1-7. doi: 10.1016/j.lungcan.2016.03.015. Epub 2016 Mar 28. PMID 27237020
- [Background] Masai K, Nakagawa K, Yoshida A, Sakurai H, Watanabe S, Asamura H, Tsuta K. Cytokeratin 19 expression in primary thoracic tumors and lymph node metastases. Lung Cancer. 2014 Dec;86(3):318-23. doi: 10.1016/j.lungcan.2014.09.018. Epub 2014 Oct 12. PMID 25453845
- [Background] Vodicka J, Mukensnabl P, Vejvodova S, Spidlen V, Kulda V, Topolcan O, Pesta M. A more sensitive detection of micrometastases of NSCLC in lymph nodes using the one-step nucleic acid amplification (OSNA) method. J Surg Oncol. 2018 Feb;117(2):163-170. doi: 10.1002/jso.24826. Epub 2017 Dec 4. PMID 29205350